CLINICAL TRIAL: NCT03056144
Title: Effect of Whole Body Vibration Therapy on Muscle Function, Gross Motor Function and Bone Mineral Density in Children With Spinal Muscular Atrophy - a Feasibility Study
Brief Title: Whole Body Vibration Therapy in Children With Spinal Muscular Atrophy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All potential participants opt to a simultaneous pharmacological clinical trial
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Manchester Metropolitan University (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Tamis Wai-mun PIN, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YBPA
Record Dates: First submitted 2016-11-08; First posted 2017-02-17 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Spinal Muscular Atrophy Type 3
Keywords: spinal muscular atrophy; total body vibration; children
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: A pilot study with a before and after study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The participants will undergo the whole body vibration therapy 1 session per day, 3 days per week for 4 weeks. The whole total whole body therapy session will last 18 minutes with 9 minutes of vibration.
  Interventions: Device: whole body vibration therapy

INTERVENTIONS:
Device: whole body vibration therapy — The whole body vibration therapy regime is as follows:
  Day Vibration 1 Rest 1 Vibration 2 Rest 2 Vibration 3 Rest 3
  1. st 1 min;12Hz 3 min 1 min;12Hz 3 min 1 min;15Hz 3 min
  2. nd 1 min;15Hz 3 min 1 min;15Hz 3 min 2 min;15Hz 3 min
  3. th 2 min;15Hz 3 min 3 min;15Hz 3 min 3 min;15Hz 3 min
  4. th 2 min;24-25Hz 3 min 2 min;24-25Hz 3 min 2 min;24-25Hz 3 min >5th 3 min;24-25Hz 3 min 3 min;24-25Hz 3 min 3 min;24-25Hz 3 min
  The participants will perform mini-squats during Vibrations 1 and 3 and weight-shifting between right and left legs during Vibration 2 on the vibration platform under the supervision of a trained research assistant.

SUMMARY:
Spinal muscular atrophy (SMA) are one of the common physical disabilities in childhood. For SMA, progressive muscle weakness and early fatigue hamper the mobility of the sufferers. Osteopenia is common for this population group due to poor bone growth and muscle disuse. As a result, non-traumatic related fractures and bone pain are common. Recently, whole body vibration therapy (WBVT) has been proven to improve bone health and muscle function in healthy adults and post-menopausal women. Among the limited studies on the WBVT for children with muscular dystrophies, promising results have been shown on gross motor function, balance, and muscle strength and the WBVT appears to be safe for children with SMA.

The present pilot study is designed to investigate if WBVT is safe and feasible for individuals with SMA and if WBVT can improve muscle function, functional abilities, postural control and bone mineral density in children with SMA. Convenience samples of 10 individuals with SMA type III will be recruited. The participants will receive the WBVT of 25 Hertz and a peak-to-peak amplitude of 4mm for a session of about 18 minutes, 3 days per week for 4 weeks. Assessment will be performed at the baseline and the completion of the intervention to examine the muscle function, functional abilities, postural control and bone mineral density of the participants.

It is anticipated that the outcomes of this pilot study for SMA may show if this intervention is safe, feasible and beneficial for children with SMA type III regarding to muscle function, functional abilities, postural control and bone mineral content and if there may be any related practical issues of this intervention to this population group. The outcomes also provide research evidence to clinicians if this intervention should be recommended to individuals of similar problems.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is an X-chromosome-linked disorder, in which there is a loss of motor neurons from the anterior horn of the spinal cord due to a deletion of the SMN1 gene. SMA is usually classified under 4 categories, based on the onset time and severity of the conditions. Type I SMA is the most severe category, when the boy is diagnosed before 6 months old and has severe muscle weakness, causing them to have poor head control and unable to sit independently. Boys with type II SMA are diagnosed between 6 to 18 months of age and able to sit independently but cannot stand or walk without any assistance. SMA type III is diagnosed between 18 months to 30 years of age and the boys can stand and walk independently but still with variable degrees of muscle weakness. Some would lose ambulation in their early adulthood and require wheelchair mobility. Type IV SMA is the mildest form with an adult onset, normal mobility and longevity. However, they also experience mild muscle weakness throughout their life. This muscle weakness would lead to early loss of ambulation, reduced pulmonary function and complications due to immobilisation such as osteoporosis. Early fatality is not uncommon.

Osteopenia due to disuse is, in fact, common in children with physical disabilities. In a study of 69 children with moderate to severe cerebral palsy (CP), it was shown that the distal femur and lumbar spine areal bone mineral density (BMD) z-scores appeared to worsen with time, which may reflect the possibility of poor bone growth velocity in individuals with CP. Fracture and bone pain are the major complications of osteopenia in CP and the majority of non-traumatic fractures occur in the femur and humerus. Other factors that may contribute to osteopenia in physical disabilities include pubertal delay, vitamin D deficiency, dietary calcium deficiency, under-nutrition and low body weight, corticosteroids or anticonvulsants. Despite of minimising these factors, osteopenia appears to persist.

Limited studies have been done to examine the bone health in children with SMA but more in children with Duchene muscular dystrophy (DMD), which have similar clinical presentations although with different pathologies. A study on 41 boys with DMD, bone density in the proximal femur was significantly decreased even in the ambulatory boys (mean z-score -1.6) and progressing rapidly to a level of 4 standard deviations below the norm when compared with normal boys. Forty-four percent of the boys had an episode of fracture, mostly in the lower limbs.

Recently whole body vibration therapy (WBVT) has been preliminarily shown as a simple and effective technique to increase bone mass, muscle mass and strength. In general, the user stands in a static position such as standing or performs some dynamic movements on a device providing vibrations from a few Hz to 50 Hz (Hertz, Hz represents the number of complete up and down movement cycle per second). It has been hypothesised that the vibrations stimulate the muscle spindles and alpha-motor neurons, eliciting a muscle contraction. The latter would increase the muscle mass and in turn, increase the bone mass. It has also been postulated that direct effect by mechanical deformation of bones and increased fluid flow in the canalicular spaces and stimulation of the osteocytes may contribute increase in bone mass with the vibration therapy. Increase in oxygen consumption, body temperature and skin blood flow (erythema) have also been demonstrated. As WBVT does not elicit a significant cardiovascular response, it appears to be safe to be used in children with various medical conditions.

In a systematic review on 22 studies (including 7 studies on CP and 2 on DMD) for the effect of WBVT on body composition and physical fitness in children and adolescents with disabilities, the authors concluded that WBVT appeared to improve bone mass and muscle strength in this population group. However, heterogeneity of the studies was noticed, including great variations in the treatment protocols and lacking of a control group and hence, no recommended minimal dosage of WBVT can be concluded. Since this review, two more randomised controlled trials (RCT) were published on children with CP. In one recent study, 30 children with spastic diplegia CP of GMFCS levels I to II were randomised into a treatment group (WBVT with traditional physiotherapy) and a control group (physiotherapy only). The treatment group received 3 lots of 3 minutes on and 3 minutes off vibration (12 to 18 Hz), 2 to 5 times per week for 3 months. Significant improvement in knee extensor strength and standing stability was reported in the treatment group. In another study in 2013, 27 children with spastic diplegia or hemiplegia CP of GMFCS levels I to III were randomised to a treatment group or control group and then crossed over after 4 weeks. The treatment group performed specific trunk exercise on the vibration platform (35 Hz), 5 to 10 minute per session, 2 to 4 sessions per week for 4 weeks. Significant improvement was found in gait speed, muscle thickness of the abdominal muscle and number of sit-ups done 1 minute. A visual improvement was also shown in sitting and standing postures.

Although it has been shown that high frequency low amplitude vibration seemed to be a safe rehabilitation in mice with muscular dystrophy, intensive strengthening exercises, which may induce more damage to the muscle fibres for children with DMD or SMA as clinically indicated with a raised serum creatine kinase (SCK) level, remain as a concern. Hence current studies on this population group targeted to examine the safety of this intervention. Three studies on children with DMD and 1 on DMD and SMA using WBVT were found. In general, it appears that WBVT seems to be safe for children with DMD or SMA. Although there might be a raised SCK level, the level would gradually reduce to the baseline level, or if not, there was no clinical sign or symptom for muscle damage. A promising result was also shown in improving bone mineral density in children with DMD. However, due to the overall small number of studies and sample sizes, there is no definite conclusion if WBVT is effective in improving the bone density and muscle strength for this population group yet.

Based on current research evidence, it has been suggested that 10 to 20 minutes per session, at least 3 times per week for minimum 26 weeks with frequency between 25 to 35 Hz and a peak to peak amplitude less than 4 mm may be an appropriate protocol targeting to improve bone mass and muscle strength of children and adolescents with disabilities. Studies of rigorous research designs and homogeneous participants are required to investigate if this recommended dosage of WBVT can improve children with disabling conditions.

Methodology This feasibility study aims to examine the safety of the WBVT on children with type III SMA. Children with type III SMA are targeted as they have adequate independence living in the community but still experience early fatigue during normal level of exercises due to the nature of their condition. They are at high risk of suffering from complications due to compromised mobility such as osteopenia, early loss of ambulation when compared with their healthy peers.

The WBVT will be performed on the GalileoTM Med L Plus (Novotech Medical GmbH) with the study participants standing with both knees flexed at least 20 degrees. The vibration frequency and duration will be increased over 5 days to the maximum of 3 minutes of 24 to 25 Hz with a peak to peak amplitude of 4mm. The participants will undergo the WBVT 1 session per day, 3 days per week for 4 weeks. The whole WBVT session will last 18 minutes with 9 minutes of vibration.

Participants:

10 children with type III SMA aged from 6 to 18 years will be recruited. The age range is extended aiming to increase the number of recruitment due to the rarity of the condition. All participants will continue their usual intervention regime, if any, during the study period.

Recruitment:

Children and families will be identified by their paediatrician at the neuromuscular clinic at the Duchess of Kent Children's Hospital in Hong Kong. Participants and/or their parents/guardians will be asked if they are interested to participate in this study and their contact details (name and contact telephone number) will be passed onto the PI. PI will contact the families by telephone.

Power analysis:

There is no previous study specifically conducted for this group of children and adolescents and hence no data is available for the power calculation. Most importantly, the aim of this study is to examine the safety and feasibility of the WBVT for this group of clients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type III spinal muscular atrophy
* Be able to stand on the vibration platform with or without support
* Be able to undertake clinical examination and DXA evaluation
* Informed consent by the participant's parent/ guardian

Exclusion Criteria:

* There is a history of fracture within 8 weeks of enrolment of the present study and acute thrombosis, muscle or tendon inflammation, renal stones, discopathy or arthritis as reported by their parent/ guardian.
* There is a history of using any of the following medications, regardless of dose, for at least 1 month, within 3 months of enrolment into the present study: anabolic agents, or growth hormone.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamis W Pin, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vry J, Schubert IJ, Semler O, Haug V, Schonau E, Kirschner J. Whole-body vibration training in children with Duchenne muscular dystrophy and spinal muscular atrophy. Eur J Paediatr Neurol. 2014 Mar;18(2):140-9. doi: 10.1016/j.ejpn.2013.09.005. Epub 2013 Oct 11. PMID 24157400
- [Background] Henderson RC, Kairalla JA, Barrington JW, Abbas A, Stevenson RD. Longitudinal changes in bone density in children and adolescents with moderate to severe cerebral palsy. J Pediatr. 2005 Jun;146(6):769-75. doi: 10.1016/j.jpeds.2005.02.024. PMID 15973316
- [Background] Stevenson RD, Conaway M, Barrington JW, Cuthill SL, Worley G, Henderson RC. Fracture rate in children with cerebral palsy. Pediatr Rehabil. 2006 Oct-Dec;9(4):396-403. doi: 10.1080/13638490600668061. PMID 17111566
- [Background] Mergler S, Evenhuis HM, Boot AM, De Man SA, Bindels-De Heus KG, Huijbers WA, Penning C. Epidemiology of low bone mineral density and fractures in children with severe cerebral palsy: a systematic review. Dev Med Child Neurol. 2009 Oct;51(10):773-8. doi: 10.1111/j.1469-8749.2009.03384.x. Epub 2009 Jul 8. PMID 19614941
- [Background] Houlihan CM, Stevenson RD. Bone density in cerebral palsy. Phys Med Rehabil Clin N Am. 2009 Aug;20(3):493-508. doi: 10.1016/j.pmr.2009.04.004. PMID 19643349
- [Background] Henderson RC, Lark RK, Gurka MJ, Worley G, Fung EB, Conaway M, Stallings VA, Stevenson RD. Bone density and metabolism in children and adolescents with moderate to severe cerebral palsy. Pediatrics. 2002 Jul;110(1 Pt 1):e5. doi: 10.1542/peds.110.1.e5. PMID 12093986
- [Background] Larson CM, Henderson RC. Bone mineral density and fractures in boys with Duchenne muscular dystrophy. J Pediatr Orthop. 2000 Jan-Feb;20(1):71-4. PMID 10641693
- [Background] Rauch F. Vibration therapy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:166-8. doi: 10.1111/j.1469-8749.2009.03418.x. PMID 19740225
- [Background] Jordan MJ, Norris SR, Smith DJ, Herzog W. Vibration training: an overview of the area, training consequences, and future considerations. J Strength Cond Res. 2005 May;19(2):459-66. doi: 10.1519/13293.1. PMID 15903391
- [Background] Rehn B, Lidstrom J, Skoglund J, Lindstrom B. Effects on leg muscular performance from whole-body vibration exercise: a systematic review. Scand J Med Sci Sports. 2007 Feb;17(1):2-11. doi: 10.1111/j.1600-0838.2006.00578.x. Epub 2006 Aug 10. PMID 16903900
- [Background] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus Mallen JA. Effect of whole-body vibration therapy on health-related physical fitness in children and adolescents with disabilities: a systematic review. J Adolesc Health. 2014 Apr;54(4):385-96. doi: 10.1016/j.jadohealth.2013.11.001. Epub 2014 Jan 1. PMID 24388109
- [Background] El-Shamy SM. Effect of whole-body vibration on muscle strength and balance in diplegic cerebral palsy: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Feb;93(2):114-21. doi: 10.1097/PHM.0b013e3182a541a4. PMID 24434887
- [Background] Unger M, Jelsma J, Stark C. Effect of a trunk-targeted intervention using vibration on posture and gait in children with spastic type cerebral palsy: a randomized control trial. Dev Neurorehabil. 2013;16(2):79-88. doi: 10.3109/17518423.2012.715313. PMID 23477461
- [Background] Novotny SA, Mader TL, Greising AG, Lin AS, Guldberg RE, Warren GL, Lowe DA. Low intensity, high frequency vibration training to improve musculoskeletal function in a mouse model of Duchenne muscular dystrophy. PLoS One. 2014 Aug 14;9(8):e104339. doi: 10.1371/journal.pone.0104339. eCollection 2014. PMID 25121503
- [Background] Chelly J, Desguerre I. Progressive muscular dystrophies. Handb Clin Neurol. 2013;113:1343-66. doi: 10.1016/B978-0-444-59565-2.00006-X. PMID 23622359
- [Background] Myers KA, Ramage B, Khan A, Mah JK. Vibration therapy tolerated in children with Duchenne muscular dystrophy: a pilot study. Pediatr Neurol. 2014 Jul;51(1):126-9. doi: 10.1016/j.pediatrneurol.2014.03.005. Epub 2014 Apr 4. PMID 24830767
- [Background] Soderpalm AC, Kroksmark AK, Magnusson P, Karlsson J, Tulinius M, Swolin-Eide D. Whole body vibration therapy in patients with Duchenne muscular dystrophy--a prospective observational study. J Musculoskelet Neuronal Interact. 2013 Mar;13(1):13-8. PMID 23445910
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823
- [Background] Mazzone E, Bianco F, Main M, van den Hauwe M, Ash M, de Vries R, Fagoaga Mata J, Stein S, De Sanctis R, D'Amico A, Palermo C, Fanelli L, Scoto MC, Mayhew A, Eagle M, Vigo M, Febrer A, Korinthenberg R, de Visser M, Bushby K, Muntoni F, Goemans N, Sormani MP, Bertini E, Pane M, Mercuri E. Six minute walk test in type III spinal muscular atrophy: a 12month longitudinal study. Neuromuscul Disord. 2013 Aug;23(8):624-8. doi: 10.1016/j.nmd.2013.06.001. Epub 2013 Jul 1. PMID 23809874
- [Background] Noto Y, Misawa S, Mori M, Kawaguchi N, Kanai K, Shibuya K, Isose S, Nasu S, Sekiguchi Y, Beppu M, Ohmori S, Nakagawa M, Kuwabara S. Prominent fatigue in spinal muscular atrophy and spinal and bulbar muscular atrophy: evidence of activity-dependent conduction block. Clin Neurophysiol. 2013 Sep;124(9):1893-8. doi: 10.1016/j.clinph.2012.12.053. Epub 2013 Apr 30. PMID 23643309
- See also: Farooq FT, Holcik M, MacKenzie A. Spinal Muscular Atrophy: Classification, Diagnosis, Background, Molecular Mechanism and Development of Therapeutics 2013. — https://www.intechopen.com/books/neurodegenerative-diseases/spinal-muscular-atrophy-classification-diagnosis-background-molecular-mechanism-and-development-of-t

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was recruited and assigned for the intervention.
Groups:
- Intervention Group: The participants will undergo the whole body vibration therapy 1 session per day, 3 days per week for 4 weeks. The whole total whole body therapy session will last 18 minutes with 9 minutes of vibration.
  whole body vibration therapy: The whole body vibration therapy regime is as follows: Day Vibration 1 Rest 1 Vibration 2 Rest 2 Vibration 3 Rest 3
  1. st 1 min;12Hz 3 min 1 min;12Hz 3 min 1 min;15Hz 3 min
  2. nd 1 min;15Hz 3 min 1 min;15Hz 3 min 2 min;15Hz 3 min
  3. th 2 min;15Hz 3 min 3 min;15Hz 3 min 3 min;15Hz 3 min
  4. th 2 min;24-25Hz 3 min 2 min;24-25Hz 3 min 2 min;24-25Hz 3 min >5th 3 min;24-25Hz 3 min 3 min;24-25Hz 3 min 3 min;24-25Hz 3 min
  The participants will perform mini-squats during Vibrations 1 and 3 and weight-shifting between right and left legs during Vibration 2 on the vibration platform under the supervision of a trained research assistant.
Period: Overall Study
Arm/Group | Intervention Group
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: no difference from the assignment in Participant flow.
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 1

OUTCOME MEASURES:

1. Primary Outcome: North Star Ambulatory Assessment
Description: examine the gross motor function of the participants. A summed score will be added from each test item.
Time Frame: 4 weeks
Reporting Status: Not Posted

2. Primary Outcome: 2-minute Walk Test
Description: assess submaximal exercise capacity by measuring the distance covered in the 2 minutes in metres
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Primary Outcome: Segmental Assessment of Trunk Control-static
Description: assess the segmental trunk control in sitting position with an ordinal score will be given in static trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
score on a scale | 8 [8 to 8]

4. Primary Outcome: Pediatric Evaluation of Disability Inventory
Description: assess functional capacities in the domains of self care, mobility and social function with a summary score in each domain. A dichotomous score will be given to each question in each domain: 0= unable and 1= able. In self care domain, there are 73 questions, i.e. maximal score is 73. In mobility domain, there are 59 questions i.e. maximal score is 59. In social function domain, there are 65 questions i.e. maximal score is 65.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
score on a scale
  PEDI- self care | 68 (0)
  PEDI- mobility | 14 (0)
  PEDI- social function | 64 (0)

5. Primary Outcome: Body Height
Description: measure height in cm
Time Frame: 4 weeks
Reporting Status: Not Posted

6. Primary Outcome: Body Weight
Description: measure weight in kilograms
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Primary Outcome: Body Mass Index
Description: calculated based on body height and weight in terms of kg/m2
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Primary Outcome: Bone Mineral Content of Femur
Description: Distal femur BMC will be measured in grams
Time Frame: 4 weeks
Reporting Status: Not Posted

9. Primary Outcome: Bone Mineral Content of Whole Body (Excluding Head)
Description: Whole body (excluding head) BMC will be measured in grams
Time Frame: 4 weeks
Reporting Status: Not Posted

10. Primary Outcome: Areal Bone Mineral Density of Femur
Description: Areal bone mineral density of femur will be measured in grams/cm2
Time Frame: 4 weeks
Reporting Status: Not Posted

11. Primary Outcome: Areal Bone Mineral Density of Total Body (Excluding Head)
Description: Areal bone mineral density of total body (excluding head) will be measured in grams/cm2
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
g/cm2 | 0.902 (0)

12. Primary Outcome: Volumetric Bone Mineral Density of Lumbar Spine
Description: Volumetric bone mineral density of lumbar spine (L2 to L4) in grams/cm3
Time Frame: 4 weeks
Reporting Status: Not Posted

13. Primary Outcome: Range of Right Hip Flexion
Description: measure hip flexion in supine using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

14. Primary Outcome: Range of Left Hip Flexion
Description: measure hip flexion in supine using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

15. Primary Outcome: Range of Right Hip Extension
Description: measure hip extension in prone using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

16. Primary Outcome: Range of Left Hip Extension
Description: measure hip extension in prone using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

17. Primary Outcome: Range of Right Hip Abduction
Description: measure hip abduction in supine using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

18. Primary Outcome: Range of Left Hip Abduction
Description: measure hip abduction in supine using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

19. Primary Outcome: Range of Right Knee Flexion
Description: measure knee flexion in prone using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

20. Primary Outcome: Range of Left Knee Flexion
Description: measure knee flexion in prone using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

21. Primary Outcome: Range of Right Knee Extension
Description: measure knee extension in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

22. Primary Outcome: Range of Left Knee Extension
Description: measure knee extension in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

23. Primary Outcome: Range of Right Ankle Dorsiflexion
Description: measure ankle dorsiflexion in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

24. Primary Outcome: Range of Left Ankle Dorsiflexion
Description: measure ankle dorsiflexion in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

25. Primary Outcome: Range of Right Ankle Plantarflexion
Description: measure ankle plantarflexion in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

26. Primary Outcome: Range of Left Ankle Plantarflexion
Description: measure ankle plantarflexion in sitting using goniometer in degrees
Time Frame: 4 weeks
Reporting Status: Not Posted

27. Primary Outcome: Muscle Strength of Right Hip Flexors
Description: measure muscle strength of hip flexors in supine using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

28. Primary Outcome: Muscle Strength of Left Hip Flexors
Description: measure muscle strength of hip flexors in supine using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

29. Primary Outcome: Muscle Strength of Right Hip Extensors
Description: measure muscle strength of hip extensors in prone using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

30. Primary Outcome: Muscle Strength of Left Hip Extensors
Description: measure muscle strength of hip extensors in prone using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

31. Primary Outcome: Muscle Strength of Right Knee Flexors
Description: measure muscle strength of knee flexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

32. Primary Outcome: Muscle Strength of Left Knee Flexors
Description: measure muscle strength of knee flexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

33. Primary Outcome: Muscle Strength of Right Knee Extensors
Description: measure muscle strength of knee extensors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

34. Primary Outcome: Muscle Strength of Left Knee Extensors
Description: measure muscle strength of knee extensors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

35. Primary Outcome: Muscle Strength of Right Hip Abductors
Description: measure muscle strength of hip abductors in supine using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

36. Primary Outcome: Muscle Strength of Left Hip Abductors
Description: measure muscle strength of hip abductors in supine using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

37. Primary Outcome: Muscle Strength of Right Ankle Dorsiflexors
Description: measure muscle strength of ankle dorsiflexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

38. Primary Outcome: Muscle Strength of Left Ankle Dorsiflexors
Description: measure muscle strength of ankle dorsiflexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

39. Primary Outcome: Muscle Strength of Right Ankle Plantarflexors
Description: measure muscle strength of ankle plantarflexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

40. Primary Outcome: Muscle Strength of Left Ankle Plantarflexors
Description: measure muscle strength of ankle plantarflexors in sitting using dynamometer in terms of Newton
Time Frame: 4 weeks
Reporting Status: Not Posted

41. Secondary Outcome: Percentage of Attendance of Participants
Description: record the percentage of attendance and comments during the intervention
Time Frame: 4 weeks
Measure: Number; unit: percentage of attendance
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
percentage of attendance | 100

42. Secondary Outcome: Visual Analogue Scale
Description: record discomfort during the intervention in a scale of 0 (no discomfort) to 10 (maximal discomfort).
Time Frame: 4 weeks
Measure: Number; unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
score on a scale | 0

43. Primary Outcome: Segmental Assessment of Trunk Control_active
Description: assess the segmental trunk control in sitting position with an ordinal score will be given in active trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
score on a scale | 8 [8 to 8]

44. Primary Outcome: Segmental Assessment of Trunk Control-reactive
Description: assess the segmental trunk control in sitting position with an ordinal score will be given in reactive trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
score on a scale | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: same definition as listed
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03056144/Prot_SAP_000.pdf